CLINICAL TRIAL: NCT04682080
Title: Comparative Evaluation of Pain Perception With a Comfort-in Jet Injection and Convantional Dental Injection in Children: a Randomized, Split-mouth, Clinical Trial
Brief Title: Pain Perception With a Comfort-ın Jet Injection and Conventional Dental Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halenur Altan, Associated Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/33
Record Dates: First submitted 2020-12-13; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Pain; Local Infiltration; Anesthesia; Fear; Anxiety; Needle Phobia
Keywords: Comfort-in jet injection system; needle-free injection; dental pain; dental anxiety and fear; color of pain
MeSH Terms: conditions — Pain; Anxiety Disorders; Toothache | interventions — Dental Health Services

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needle-free injection group (Active Comparator): In needle-free injection techniques, 4% articaine with 1/100.000 epinephrine (Ultracaine DS forte) was injected using the Comfort-In system. Pain intensity and anxiety levels of patients were measured.
  Interventions: Behavioral: Needle-free injection
- Dental injection group (Active Comparator): In the conventional dental-injection method, 4% articaine with 1/100.000 epinephrine (Ultracaine DS forte) was injected using a 27G, 50-mm, disposable syringe with a needle. Pain intensity and anxiety levels of patients were measured.
  Interventions: Behavioral: Needle-free injection

INTERVENTIONS:
Behavioral: Needle-free injection — This study was performed among children aged 4-10 years who required dental treatment and were treated at the Department of Pedodontics, Faculty of Dentistry, Gaziosmanpasa University. A total of 120 patients were evaluated in accordance with the exclusion criteria and 94 children (39 girls and 55 boys) were included in this study. Children who needed dental treatment were randomly divided into two groups. All dental injections were administered by the same operator (MB), a pediatric dentist with two years of experience in using the Comfort-In system.
  In both groups, the children were asked to rate their pain intensity by choosing the closest statement on the colorful Wong-Baker Pain Scale at four time points: immediately after injection (Pain 1), during treatment (Pain 2), at the end of the treatment (Pain 3) and postoperative first day.Anxiety levels were recorded using the Modified Children's Dental Anxiety Scale face version
  Other Names: Dental injection

SUMMARY:
The investigators aimed to compare the effectiveness of the Comfort-in system, which is a jet injection type, and infiltrative anesthesia with a traditional injector, and to measure the effect of children's anxiety on the severity of pain.

DETAILED DESCRIPTION:
Among the children between the ages of 4 and 10 who were admitted to clinic between 2018-2020, whose clinical and radiographic examinations were completed; Patients with deciduous teeth that needed the same dental treatment (filling or amputation) with symmetrical local anesthesia application and positive (3) or definitely positive (4) according to the Frankl Behavior Evaluation Scale were included in the study. In study with a split-mouth design, infiltration anesthesia was applied with a conventional dental injector to one of the symmetrical teeth requiring the same treatment, while the Comfort-in jet injection system was applied to the other by the same physician. Patients were randomized into two grups according to the injection technique.

Group1: Needle-free injection system(Comofrt-In) 2:Dental injection method. The pain intensity was assessed during anesthesia(Pain 1), during treatment(Pain 2), at the end of the treatment(Pain 3) and on the postoperative 1st day (Pain 4)by the specially 7 colors (white, yellow, green, blue, magenta, red, black) using the Wong-Baker facial expressions and pain grading scale.Anxiety levels were recorded using the Modified Children's Dental Anxiety Scale face version.

The data were analyzed by IBM SPSS Statistics 19, the significance level was taken as p <0.05.The datas were analyzed with a three-way variance method in repeated.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 4-10 years
* Having no developmental or systemic disorder or no history of allergy
* Having "positive" or "definitely positive" cooperation level according to the Frankl Behavior Scale
* Having sufficient mouth opening
* Operation only on primary teeth
* Having decayed teeth that require anesthesia

Exclusion Criteria:

* Patients younger than four years, older than 10 years,
* Patients with systemic or developmental disorders
* Children with an allergy history
* 'Negative' or 'definitly negative' behavior rating according to the Frankl scale
* Patients whose mouth opening is not sufficient for dental treatment
* Operating only on permanent teeth
* Teeth that are beyond the treatment stage
* When pain occurred during treatment, supplemental anesthetics administrated, and these children were excluded.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Pain at different anesthesia methods | after dental treatments to 24 hour
  The pain perception scores in the two anesthesia methods were assessed with Wong-Baker Pain Scale (Wong-Baker Scale is pain assessment method.It consists of 6 facial expressions that are evaluated from 0 to 10 according to the severity of the pain. Values between 0-4 indicate mild pain, values between 4-6 indicate moderate pain, values between 6-8 indicate severe pain and values between 8-10 indicate unbearable pain).
Anxiety level of children | after dental treatments(40 minutes)
  Anxiety level of children were assesed with Modified Child Dental Anxiety Scale (Modified Child Dental Anxiety Scale is anxiety assessment method. It consist of 8 questions about dental procedures. Each questions are evaluated 5 faces from smiles to cries according to the severity of tne anxiety. Patients with a Modified Child Dental Anxiety Scale value below 26 have less anxiety, and patients with a value of 26 and above have a high level of anxiety.
Color of pain during anesthesia. | immediately after injection(2 minutes),
  The pain perception scores in the two anesthesia methods were assessed with 7 colorful (white,yellow, green, blue, purple, red and black) Wong-Baker Pain Scale (Wong-Baker Scale is pain assessment method.It consists of 6 facial expressions that are evaluated from 0 to 10 according to the severity of the pain. Values between 0-4 indicate mild pain, values between 4-6 indicate moderate pain, values between 6-8 indicate severe pain and values between 8-10 indicate unbearable pain)
Children's preferred anesthesia method | After using each dental injection method(2 weeks).
  Children's preferred anesthesia method was asked for children after two different injection tecniques used.

CONTACTS AND LOCATIONS:
Overall Officials: Halenur Altan, Assoc Prof., Principal Investigator — Tokat Gaziosmanpasa University, Faculty of Dentistry, Department of Pediatric Dentistry
Locations (1):
- Tokat Gaziosmanpasa University, Faculty of Dentistry, Tokat Province, Center, Turkey (Türkiye)

REFERENCES:
- [Background] Altan H, Cevik H, Dogru S, Cosgun A, Suren M, Okan I. The pain colour of children with toothache in Turkish population. BMC Oral Health. 2019 Apr 18;19(1):59. doi: 10.1186/s12903-019-0756-y. PMID 30999904
- [Background] Arapostathis KN, Dabarakis NN, Coolidge T, Tsirlis A, Kotsanos N. Comparison of acceptance, preference, and efficacy between jet injection INJEX and local infiltration anesthesia in 6 to 11 year old dental patients. Anesth Prog. 2010 Spring;57(1):3-12. doi: 10.2344/0003-3006-57.1.3. PMID 20331333
- [Background] Oliveira ACA, Amorim KS, Nascimento Junior EMD, Duarte ACB, Groppo FC, Takeshita WM, Souza LMA. Assessment of anesthetic properties and pain during needleless jet injection anesthesia: a randomized clinical trial. J Appl Oral Sci. 2019 Jan 14;27:e20180195. doi: 10.1590/1678-7757-2018-0195. PMID 30673030
- [Background] Armfield JM. Development and psychometric evaluation of the Index of Dental Anxiety and Fear (IDAF-4C+). Psychol Assess. 2010 Jun;22(2):279-87. doi: 10.1037/a0018678. PMID 20528055
- [Background] Burkitt E, Barrett M, Davis A. Children's colour choices for completing drawings of affectively characterised topics. J Child Psychol Psychiatry. 2003 Mar;44(3):445-55. doi: 10.1111/1469-7610.00134. PMID 12635973
- [Background] Howard KE, Freeman R. Reliability and validity of a faces version of the Modified Child Dental Anxiety Scale. Int J Paediatr Dent. 2007 Jul;17(4):281-8. doi: 10.1111/j.1365-263X.2007.00830.x. PMID 17559456
- [Background] Khatri A, Kalra N. A comparison of two pain scales in the assessment of dental pain in East delhi children. ISRN Dent. 2012;2012:247351. doi: 10.5402/2012/247351. Epub 2012 Feb 14. PMID 22461986
- [Background] Langthasa M, Yeluri R, Jain AA, Munshi AK. Comparison of the pain perception in children using comfort control syringe and a conventional injection technique during pediatric dental procedures. J Indian Soc Pedod Prev Dent. 2012 Oct-Dec;30(4):323-8. doi: 10.4103/0970-4388.108931. PMID 23514685
- [Background] Makade CS, Shenoi PR, Gunwal MK. Comparison of acceptance, preference and efficacy between pressure anesthesia and classical needle infiltration anesthesia for dental restorative procedures in adult patients. J Conserv Dent. 2014 Mar;17(2):169-74. doi: 10.4103/0972-0707.128063. PMID 24778516
- [Background] Ocak H, Akkoyun EF, Colpak HA, Demetoglu U, Yucesoy T, Kilic E, Alkan A. Is the jet injection effective for teeth extraction? J Stomatol Oral Maxillofac Surg. 2020 Feb;121(1):19-24. doi: 10.1016/j.jormas.2019.05.001. Epub 2019 May 8. PMID 31077857
- [Background] Munshi AK, Hegde A, Bashir N. Clinical evaluation of the efficacy of anesthesia and patient preference using the needle-less jet syringe in pediatric dental practice. J Clin Pediatr Dent. 2001 Winter;25(2):131-6. doi: 10.17796/jcpd.25.2.q6426p853266q575. PMID 11314212
- [Background] Saravia ME, Bush JP. The needleless syringe: efficacy of anesthesia and patient preference in child dental patients. J Clin Pediatr Dent. 1991 Winter;15(2):109-12. PMID 1931745
- [Background] Sermet Elbay U, Elbay M, Yildirim S, Kaya E, Kaya C, Ugurluel C, BaydemIr C. Evaluation of the injection pain with the use of DentalVibe injection system during supraperiosteal anaesthesia in children: a randomised clinical trial. Int J Paediatr Dent. 2016 Sep;26(5):336-45. doi: 10.1111/ipd.12204. Epub 2015 Sep 15. PMID 26369274
- [Background] Wogelius P, Poulsen S, Sorensen HT. Prevalence of dental anxiety and behavior management problems among six to eight years old Danish children. Acta Odontol Scand. 2003 Jun;61(3):178-83. doi: 10.1080/00016350310003468. PMID 12868693